CLINICAL TRIAL: NCT01141790
Title: Analysis of Vital, Facial and Muscular Responses Front to Music or Message in Coma, Vegetative State or Sedated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Masking: Single | Purpose: Supportive Care
Other Study IDs: FAPESP 06/61338-5
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Consciousness Disorders; Communication; Intensive Care
Keywords: Glasgow Coma Scale; Glasgow Outcome Scale; Ethics
MeSH Terms: conditions — Consciousness Disorders; Communication

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Silence (Placebo Comparator): The control group listened "silence" and was evaluated the same things.
  Interventions: Other: Music and voice message

INTERVENTIONS:
Other: Music and voice message

SUMMARY:
Objectives: (1) To check music or voice message influence on vital signs, facial expressions or muscular tonus of coma, vegetative or sedated patients; (2) To connect the existence of patient's responsiveness with the Glasgow Coma Scale or with the Ramsay Sedation Scale; (3)To evaluate the relation between the response and the score of Glasgow Outcome Scale.

ELIGIBILITY:
Inclusion Criteria:

* To be in disorder of consciousness;
* To be evaluated according to one of the Scales and to have a score in the study range: in physiological comas, score between 3 to 8 Glasgow Coma Scale (GCS); in induced coma, one of the last two scores of Ramsay Sedation Scale (RSS), R5 or R6;
* To have hearing function preserved according to family;
* To have written consent from the family or responsible party for the patient's participation

Exclusion Criteria:

* Score between 9 to 15 in GCS or scores R1, R2, R3 or R4 in RSS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- HCFMUSP - Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: website of principal investigator — http://claudiapuggina@usp.br